CLINICAL TRIAL: NCT03661320
Title: A Phase 3, Randomized, Study of Neoadjuvant Chemotherapy Alone Versus Neoadjuvant Chemotherapy Plus Nivolumab or Nivolumab and BMS-986205, Followed by Continued Post- Surgery Therapy With Nivolumab or Nivolumab and BMS-986205 in Participants With Muscle- Invasive Bladder Cancer
Brief Title: A Study to Compare Chemotherapy Alone Versus Chemotherapy Plus Nivolumab or Nivolumab and BMS-986205, Followed by Continued Therapy After Surgery With Nivolumab or Nivolumab and BMS-986205 in Participants With Muscle Invasive Bladder Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA017-078; 2024-512158-12 (Other: EU CT Number)
Record Dates: First submitted 2018-09-05; First posted 2018-09-07 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Urinary Bladder Neoplasms; Muscle-Invasive Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Nivolumab; Gemcitabine; Drug Therapy; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Gemcitabine/Cisplatin (GC) Chemotherapy (Active Comparator)
  Interventions: Drug: Gemcitabine; Drug: Cisplatin
- Arm B: Nivolumab + GC Chemotherapy (Experimental)
  Interventions: Biological: Nivolumab; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Biological: Nivolumab — Specified dose on specified days
  Other Names: Opdivo; BMS-936558
  Arms: Arm B: Nivolumab + GC Chemotherapy
Drug: Gemcitabine — Specified dose on specified days
  Other Names: Chemotherapy
Drug: Cisplatin — Specified dose on specified days
  Other Names: Chemotherapy

SUMMARY:
The purpose of this study is to compare nivolumab plus neoadjuvant gemcitabine/cisplatin (GC) chemotherapy, followed by post-surgery continuation of immuno-oncology (IO) therapy, with neoadjuvant GC chemotherapy alone in adult participants with previously untreated muscle-invasive bladder cancer (MIBC).

ELIGIBILITY:
Inclusion Criteria:

* Participant must be deemed eligible for Radial Cystectomy (RC) by his/her oncologist and/or urologist, and must agree to undergo Radial Cystectomy (RC) after completion of neoadjuvant therapy.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1

Exclusion Criteria:

* Clinical evidence of positive lymph node(s) (LN) (≥ 10 mm in short axis) or metastatic bladder cancer
* Prior systemic therapy, radiation therapy, or surgery for bladder cancer other than trans urethral resection of bladder tumor (TURBT) or biopsies is also not permitted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 855 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2026-02-16 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) rate, in all randomized participants | Approximately 43 months
  Arm B vs. Arm A
Event-Free Survival (EFS), in all randomized participants | Approximately 36 months
  Arm B vs. Arm A

SECONDARY OUTCOMES:
Overall Survival (OS) in all randomized participants | Approximately 60 months
  Arm B vs. Arm A
Incidence of Adverse Events (AE) in participants who received at least one treatment dose | Approximately 60 months
Incidence of Serious Adverse Events (SAE) in participants who received at least one treatment dose | Approximately 60 months
Incidence of deaths in participants who received at least one treatment dose | Approximately 60 months
Incidence of laboratory abnormalities in participants who received at least one treatment dose | Approximately 60 months
pCR rate, descriptively in all concurrently randomized participants | Approximately 43 months
  Arm C vs. Arm B and Arm A
EFS, descriptively in all concurrently randomized participants | Approximately 36 months
  Arm C vs. Arm B and Arm A
OS, descriptively in all concurrently randomized participants | Approximately 60 months
  Arm C vs. Arm B and Arm A

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (171):
- United States (26):
  - Local Institution - 0022, Tucson, Arizona
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - Local Institution - 0021, Littleton, Colorado
  - Local Institution - 0036, Pensacola, Florida
  - Local Institution - 0004, Tampa, Florida
  - Local Institution - 0144, Atlanta, Georgia
  - Local Institution - 0005, Chicago, Illinois
  - Local Institution - 0006, Peoria, Illinois
  - Local Institution - 0181, Columbia, Maryland
  - Local Institution - 0009, Boston, Massachusetts
  - Local Institution - 0166, Boston, Massachusetts
  - Local Institution - 0209, Boston, Massachusetts
  - Local Institution - 0025, Minneapolis, Minnesota
  - Local Institution - 0129, Minneapolis, Minnesota
  - Local Institution - 0183, Omaha, Nebraska
  - Local Institution - 0001, Omaha, Nebraska
  - Local Institution - 0024, Las Vegas, Nevada
  - Local Institution - 0029, Albany, New York
  - Local Institution - 0069, Lake Success, New York
  - Local Institution - 0047, New York, New York
  - Local Institution - 0191, Cleveland, Ohio
  - Local Institution - 0028, Tigard, Oregon
  - Local Institution - 0189, Charleston, South Carolina
  - Local Institution - 0007, Nashville, Tennessee
  - Local Institution - 0030, Austin, Texas
  - Local Institution - 0023, Norfolk, Virginia
- Argentina (3):
  - Local Institution - 0051, Capital Federal, Buenos Aires
  - Local Institution - 0049, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Local Institution - 0151, Ciudad Autonoma Buenos Aires, Distrito Federal
- Australia (7):
  - Local Institution - 0131, Garran, Australian Capital Territory
  - Local Institution - 0130, Kingswood, New South Wales
  - Local Institution - 0157, Macquarie University, New South Wales
  - Local Institution - 0043, St Leonards, New South Wales
  - Local Institution - 0143, North Adelaide, South Australia
  - Local Institution - 0037, Heidelberg, Victoria
  - Local Institution - 0038, Murdoch, Western Australia
- Austria (4):
  - Local Institution - 0090, Klagenfurt
  - Local Institution - 0091, Krems
  - Local Institution - 0011, Linz
  - Local Institution - 0012, Vienna
- Belgium (3):
  - Local Institution - 0060, Brussels
  - Local Institution - 0063, Ghent
  - Local Institution - 0062, Wilrijk
- Brazil (10):
  - Local Institution - 0094, Fortaleza, Ceará
  - Local Institution - 0099, Ipatinga, Minas Gerais
  - Local Institution - 0092, Ijuí, Rio Grande do Sul
  - Local Institution - 0212, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0097, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0098, Barretos, São Paulo
  - Local Institution - 0095, Jaú, São Paulo
  - Local Institution - 0093, São José do Rio Preto, São Paulo
  - Local Institution - 0164, Rio de Janeiro
  - Local Institution - 0214, São Paulo
- Canada (4):
  - Local Institution - 0159, Kelowna, British Columbia
  - Local Institution - 0182, North York, Ontario
  - Local Institution - 0192, Chicoutimi, Quebec
  - Local Institution - 0190, Montreal, Quebec
- Chile (4):
  - Local Institution - 0053, Santiago, Santiago Metropolitan
  - Local Institution - 0052, Santiago, Santiago Metropolitan
  - Local Institution - 0210, Santiago, Santiago Metropolitan
  - Local Institution - 0054, Santiago, Santiago Metropolitan
- Colombia (3):
  - Local Institution - 0201, Colombia, Bogota D.C.
  - Local Institution - 0104, Bucaramanga
  - Local Institution - 0103, Montería
- Finland (3):
  - Local Institution - 0148, Helsinki
  - Local Institution - 0145, Tampere
  - Local Institution - 0146, Turku
- France (16):
  - Local Institution - 0202, Brest, Finistère
  - Local Institution - 0204, Créteil, Val-de-Marne
  - Local Institution - 0205, Amiens
  - Local Institution - 0198, Angers
  - Local Institution - 0101, Besançon
  - Local Institution - 0217, Bordeaux
  - Local Institution - 0199, Clermont-Ferrand
  - Local Institution - 0206, La Tronche
  - Local Institution - 0075, Marseille
  - Local Institution - 0200, Montpellier
  - Local Institution - 0074, Nice
  - Local Institution - 0163, Paris
  - Local Institution - 0020, Pierre Benite Cedax
  - Local Institution - 0188, Saint-Herblain
  - Local Institution - 0002, Strasbourg
  - Local Institution - 0003, Toulouse
- Germany (13):
  - Local Institution - 0100, Mainz, Rhineland-Palatinate
  - Local Institution - 0078, Aachen
  - Local Institution - 0015, Erfurt
  - Local Institution - 0081, Essen
  - Local Institution - 0086, Frankfurt am Main
  - Local Institution - 0080, Göttingen
  - Local Institution - 0013, Herne
  - Local Institution - 0010, Jena
  - Local Institution - 0084, Lübeck
  - Local Institution - 0079, Magdeburg
  - Local Institution - 0082, München
  - Local Institution - 0016, Nuremberg
  - Local Institution - 0085, Trier
- Greece (3):
  - Local Institution - 0195, Athens, Attikí
  - Local Institution - 0031, Larissa, Thessalía
  - Local Institution - 0194, Chaïdári
- Israel (4):
  - Local Institution - 0196, Tel Aviv, Tel Aviv
  - Local Institution - 0068, Beersheba
  - Local Institution - 0066, Haifa
  - Local Institution - 0067, Ramat Gan
- Italy (7):
  - Local Institution - 0064, Bari
  - Local Institution - 0193, Meldola (FC)
  - Local Institution - 0032, Milan
  - Local Institution - 0065, Modena
  - Local Institution - 0033, Padua
  - Local Institution - 0034, Pisa
  - Local Institution - 0035, Roma
- Japan (16):
  - Local Institution - 0186, Komaki, Aichi-ken
  - Local Institution - 0184, Sapporo, Hokkaido
  - Local Institution - 0177, Sapporo, Hokkaido
  - Local Institution - 0185, Sapporo, Hokkaido
  - Local Institution - 0179, Tsukuba, Ibaraki
  - Local Institution - 0171, Kita-gun, Kagawa-ken
  - Local Institution - 0169, Yokohama, Kanagawa
  - Local Institution - 0168, Niigata, Niigata
  - Local Institution - 0173, Sayama, Osaka
  - Local Institution - 0175, Takatsuki, Osaka
  - Local Institution - 0176, Hidaka-shi, Saitama
  - Local Institution - 0170, Hamamatasu, Shizuoka
  - Local Institution - 0178, Minato-ku, Tokyo
  - Local Institution - 0172, Shinjuku-ku, Tokyo
  - Local Institution - 0174, Fukuoka
  - Local Institution - 0180, Kyoto
- Mexico (4):
  - Local Institution - 0160, La Paz, BAJA Californa SUR
  - Local Institution - 0102, Zapopan, Jalisco
  - Local Institution - 0056, Monterrey, Nuevo León
  - Local Institution - 0105, Colima
- Netherlands (3):
  - Local Institution - 0070, Amsterdam
  - Local Institution - 0072, Groningen
  - Local Institution - 0073, Sittard-Geleen
- New Zealand (2):
  - Local Institution - 0087, Auckland
  - Local Institution - 0089, Christchurch
- Norway (3):
  - Local Institution - 0158, Grålum
  - Local Institution - 0132, Lorenskog
  - Local Institution - 0133, Oslo
- Portugal (2):
  - Local Institution - 0153, Lisbon
  - Local Institution - 0152, Porto
- Romania (3):
  - Local Institution - 0219, Cluj-Napoca
  - Local Institution - 0076, Craiova
  - Local Institution - 0058, Sector 2
- Local Institution, Saint Petersburg, Russia
- Local Institution - 0154, Singapore, Singapore
- South Korea (10):
  - Local Institution - 0137, Goyang-si, Gyeonggi-do
  - Local Institution - 0203, Seongnam-si, Kyǒnggi-do
  - Local Institution - 0220, Busan
  - Local Institution - 0218, Daegu
  - Local Institution - 0208, Gyeongsangnam-do
  - Local Institution - 0215, Seongnam-si
  - Local Institution - 0140, Seoul
  - Local Institution - 0136, Seoul
  - Local Institution - 0211, Seoul
  - Local Institution - 0138, Seoul
- Spain (6):
  - Local Institution - 0113, Lugo
  - Local Institution - 0111, Madrid
  - Local Institution - 0112, Madrid
  - Local Institution - 0114, Madrid
  - Local Institution - 0156, Málaga
  - Local Institution - 0109, Seville
- Taiwan (4):
  - Local Institution - 0135, Kaohsiung City
  - Local Institution - 0165, Taichung
  - Local Institution - 0141, Taipei
  - Local Institution - 0139, Taipei
- United Kingdom (6):
  - Local Institution - 0128, Chelmsford, Essex
  - Local Institution - 0127, York, Yorkshire
  - Local Institution - 0122, Glasgow
  - Local Institution - 0117, Lancaster
  - Local Institution - 0121, London
  - Local Institution - 0124, Oxford

REFERENCES:
- [Derived] Grivas P, Koshkin VS, Chu X, Cole S, Jain RK, Dreicer R, Cetnar JP, Sundi D, Gartrell BA, Galsky MD, Woo B, Li-Ning-Tapia E, Hahn NM, Carducci MA. PrECOG PrE0807: A Phase 1b Feasibility Trial of Neoadjuvant Nivolumab Without and with Lirilumab in Patients with Muscle-invasive Bladder Cancer Ineligible for or Refusing Cisplatin-based Neoadjuvant Chemotherapy. Eur Urol Oncol. 2024 Aug;7(4):914-922. doi: 10.1016/j.euo.2023.11.022. Epub 2023 Dec 27. PMID 38155060
- [Derived] Sonpavde G, Necchi A, Gupta S, Steinberg GD, Gschwend JE, Van Der Heijden MS, Garzon N, Ibrahim M, Raybold B, Liaw D, Rutstein M, Galsky MD. ENERGIZE: a Phase III study of neoadjuvant chemotherapy alone or with nivolumab with/without linrodostat mesylate for muscle-invasive bladder cancer. Future Oncol. 2020 Jan;16(2):4359-4368. doi: 10.2217/fon-2019-0611. Epub 2019 Dec 11. PMID 31823654
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT03661320.html